CLINICAL TRIAL: NCT06502314
Title: The Effectiveness of Stress Management Training Given to First-class Health Students in Perceiving and Coping With Stress and Developing Resilience: A Randomized Controlled Trial
Brief Title: The Effectiveness of Stress Management Training on Perceiving and Coping With Stress and Developing Resilience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Sercan, Assistant Professor, Kutahya Health Sciences University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: KHSU-MANSUROGLU-001
Record Dates: First submitted 2024-07-08; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Stress Management; Perceived Stress; Coping Strategy; Psychological Resilience
Keywords: Perceived stress; stress management; psychological resilience; health students; mental health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): In the first interview with the students assigned to the intervention group, students were informed about the purpose of the study and the process, and pre-tests were applied to the students after their consent was obtained. After 1 week, students randomly assigned to the intervention group were given psychoeducation on stress management consisting of 7 modules each lasting 120 minutes (with a break), on a day determined during the week for 7 weeks. Two weeks after the training was completed, post-tests were applied to the intervention group students.
  Interventions: Behavioral: Stress management training
- control group (No Intervention): In the first interview with the students assigned to the control group, students were informed about the purpose of the study and the process, and pre-tests were applied to the students after their consent was obtained. Ten weeks after, post-tests were applied to the control group students. During this process, no intervention was applied to the control group. After the study was completed, the same stress management training was given to the control group.

INTERVENTIONS:
Behavioral: Stress management training — It is a psychoeducational program that includes seven modules (1. Stress and its components, 2. Stress Management, 3. Crisis and its components, 4. Crisis Management, 5. Anger and its components, 6. Anger Management, 7. Psychological resilience)
  .
  Arms: intervention group

SUMMARY:
Associate degree students studying in the field of health perform their professions in the status of intermediate staff related to health in our country. They are in direct or indirect contact with every segment of the society within the health system. They are also in a multidisciplinary team. This enables them to interact within the team. Therefore, it can be clearly said that the stress they will be in may affect other team members. In previous studies in the literature, it is seen that more studies have been conducted with undergraduate health professional candidates. However, considering that associate degree health students start their professional life at a younger age, it can be thought that they may have more difficulties in coping with the stress that the health sector may cause. This situation can be facilitated by strengthening their psychological resilience. In this study, it can be said that it is important to provide stress management training and measure its effectiveness by taking these factors into consideration. It can be thought that the results will contribute to the importance by filling the gap in the literature.

Objective: This study was a pretest-posttest randomised controlled psychoeducational intervention in which the effect of stress management training given to first-year health students on their perceived stress, coping methods and psychological resilience was examined.

Research hypotheses H1: Perceived stress post-test scores of first-year health students who received stress management training will be lower than those who did not receive the same training.

H2: The post-test scores of the first-year health students who received stress management training will be higher than the post-test scores of the students who did not receive the same training.

H3: First-year health students who receive stress management training will have higher psychological resilience post-test scores than students who do not receive the same training.

Methods: The study was conducted with 102 health students, 51 intervention and 51 control. Randomly assigned intervention group received stress management training consisting of 7 modules for 7 weeks. No intervention was given to the control group. Data were collected using sociodemographic form, perceived stress scale, stress coping methods scale and short psychological resilience scale. Pre-test and post-tests were administered to both groups.

DETAILED DESCRIPTION:
This study, which examined the effect of stress management training given to health students on students' perceived stress, coping methods with stress and psychological resilience. The population of this pretest-posttest randomised controlled study consisted of 126 first-year health students studying in the associate degree departments of the central vocational school of a health university in western Turkey. The sample consisted of students who met the inclusion criteria and voluntarily accepted to participate in the study. The study was completed with 102 students, 51 intervention-51 control. First-year associate degree health students who voluntarily accepted to participate in the study, who were 18 years of age or older, and who were continuing their active education were included in the study. Students who did not meet the specified inclusion criteria were excluded from the study. The students participating in the study were not informed which group they were in. Single blinding method was used in the study because the researcher was involved in group allocation, intervention and data collection tasks. A total of 126 first-year students studying at a vocational school were evaluated by the researcher according to the inclusion or exclusion criteria. As a result, 102 participants were randomised and assigned to the intervention and control groups. In order to reduce selection bias in determining the intervention and control groups, the individuals to be included in the sample were determined using the www.random.org website. The dependent variables of the study are perceived stress scale, coping methods with stress scale and short psychological resilience scale. Stress management training is the independent variable. Sociodemographic data of the students were the control variable of the study. In this face-to-face study, students who met the inclusion criteria were randomised and assigned to the groups. In the first interview with the students assigned to the intervention and control groups, students were informed about the purpose of the study and the process, and pre-tests were applied to the students after their consent was obtained. After 1 week, students randomly assigned to the intervention group were given psychoeducation on stress management consisting of 7 modules each lasting 120 minutes (with a break), on a day determined during the week for 7 weeks. Stress management training was given by the researcher, who has a master's degree in Community Mental Health Nursing and a doctoral degree in Mental Health and Psychiatric Nursing and has received training on stress and coping with stress. Two weeks after the training was completed, post-tests were applied to the intervention and control group students. During this process, no intervention was applied to the control group. After the study was completed, the same stress management training was given to the control group. For the scales used in the study, permission was obtained from the authors who developed the scales and conducted the adaptation studies into Turkish. Written permission was obtained from the ethics committee of the university where the study was conducted (number 2024/03-04 on 05.03.2024) for ethical compliance and implementation. Informed consent was obtained after explaining the purpose of the study to the students participating in the study. In addition, the ethical principles of the current Helsinki Declaration were adhered to during the study. In this study, firstly, power analysis was performed to determine the sample size. Mean and standard deviation were used as descriptive statistics for quantitative variables determined by measurement, and number and percentage were used as descriptive statistics for qualitative variables determined by counting. Chi-square test and Fisher's exact test were used to analyse the similarity of the groups. After the normality analyses showed that the data had a normal distribution, independent sample t test and dependent sample t test were used for comparisons of pre-test and post-test scores within and between groups. Analysis of covariance (ANCOVA) was used to determine the effectiveness level of psychoeducation. In order to determine the effect size, Eta Squared (µ²) values were taken into consideration and these values were interpreted by taking the values determined by Cohen as criteria (small if .01, medium if .06 and above, and large if .14 and above). Cronbach's Alpha was calculated for reliability analysis. Analyses were performed with Statistical Package for the Social Sciences version 25 and p<0.05 was considered statistically significant in comparisons.

ELIGIBILITY:
Inclusion Criteria:

* First-year associate degree health students who voluntarily accepted to participate in the study,
* Who were 18 years of age or older,
* Who were continuing their active education.

Exclusion Criteria:

* First-year associate degree health students who voluntarily not accepted to participate in the study,
* Who were under 18 years of age,
* Who were not continuing their active education.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2024-03-06 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
Change in "Perceived Stress Scale" scores | It was applied as a pre-test before the intervention and as a post-test 2 weeks after the intervention completed, within 1 week, and the change was observed.
  This scale evaluates the stress perceptions of individuals in the face of certain situations encountered in their lives. The scale has a five-point Likert scale. The scale has two sub-dimensions but the total scale score was used for this study. The lowest score that can be obtained from the scale is 0 and the highest score is 56. The higher the score obtained by the individuals from the scale, the higher the stress perception. It was aimed to compare and evaluate the change in perceived stress levels of the participants before and after the planned psychoeducation for 7 weeks.
Change in "Stress Coping Methods Scale" scores | It was applied as a pre-test before the intervention and as a post-test 2 weeks after the intervention completed, within 1 week, and the change was observed.
  The coping methods scale was used to measure coping methods with stress. The scale consists of a five-factor structure but the total scale score was used for this study. Consisting of 24 statements, the scale is graded in 5-point Likert type. It can be said that individuals develop methods of coping with stress as the score they get from the scale increases. It was aimed to compare and evaluate the changes in the participants' methods of coping with stress before and after the psychoeducation planned for 7 weeks.
Change in "Brief Resilience Scale" scores | It was applied as a pre-test before the intervention and as a post-test 2 weeks after the intervention completed, within 1 week, and the change was observed.
  The scale is a 5-point Likert-type, 6-item, self-report measurement tool developed in order to measure the psychological resilience of individuals. High scores indicate high psychological resilience. It was aimed to compare and evaluate the changes in the participants' psychological resilience before and after the psychoeducation planned for 7 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Sercan Mansuroğlu, PhD, Study Director — Kutahya Health Sciences University
Locations (1):
- Kutahya Health Sciences University, Kütahya, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-08): https://cdn.clinicaltrials.gov/large-docs/14/NCT06502314/Prot_SAP_000.pdf